CLINICAL TRIAL: NCT03777306
Title: The Myeloma Pack: A Multi-Modality Educational Intervention Strategy to Engage Patients With Multiple Myeloma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Smith Giri, PI, University of Alabama at Birmingham
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-300000121
Record Dates: First submitted 2018-09-27; First posted 2018-12-17 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Multiple Myeloma
Keywords: Educational intervention
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Multi-modality didactic education program implemented in parallel to standard cancer treatment to improve QoL for patients with MM
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM A EARLY INTERVENTION GROUP (Experimental): In Arm A, the intervention group, the participants will start on the program immediately. The participants will receive MPI educational program, implemented in parallel with standard of care treatment. The MPI is implemented at the time of enrollment x 12 weeks
  Interventions: Other: ARM A EARLY INTERVENTION GROUP
- ARM B DELAYED INTERVENTION GROUP (Experimental): Arm B, is a wait-list control group that will serve as the control. The wait-list control group will be observed for an initial 12 week period while receiving usual care and then have the educational intervention implemented from week 12-24 in parallel with standard of care
  Interventions: Other: ARM B DELAYED INTERVENTION GROUP

INTERVENTIONS:
Other: ARM A EARLY INTERVENTION GROUP — Post randomization, all patients will take baseline survey to assess their level of stress prior to starting the educational program During the educational interventions they will receive
  * 1 video/picture/worksheet per week covering the topic to be covered.
  * 1 phone/week by the Health Advisor, to discuss the topic for the week s/as their disease, stress and anxiety management, life organization, adherence skills, healthy eating and sleeping). Participant and the health advisor will also set up a "Tiny Step"" to serve as a goal for the week .
  * 3 emails/texts through the week, to remind about the topic covered, or to encourage them on their Tiny Step goal.
  After 12 weeks on the program participants will re-take the surveys to assess the level of stress.
  Arms: ARM A EARLY INTERVENTION GROUP
Other: ARM B DELAYED INTERVENTION GROUP — The educational intervention is similar as in ARM A except that the participants will receive standard of care for the first 12 weeks post randomization and then begin the educational intervention
  Arms: ARM B DELAYED INTERVENTION GROUP

SUMMARY:
Multiple Myeloma (MM) patients are prone to poor quality of life (QoL) as a result of the anxiety and depression they suffer due to a poor understanding of their disease. Improving patient understanding of their illness and addressing issues that induce distress impacts QoL. This prospective, interventional study is designed to see if a structured psycho-educational program called "the myeloma pack intervention" (MPI), implemented in parallel with standard cancer treatment, can improve QoL for patients with MM.

DETAILED DESCRIPTION:
The purpose of this research study is to see if the MPI educational program, implemented in parallel with standard of care treatment, can improve overall quality of life (QoL) for MM patients. This program will be delivered to the study participants by multiple modes of communication including written material in a boxed pack, online tutorials, telephone and text message follow up. If they do not have online access at home, the study coordinators will arrange access for the participants at the Clinic. A health advisor will work with the physicians to coordinate their participation in the program while they are on active treatment for myeloma. The Pack Health Advisors will only give them guidance about the study and they will not provide any kind of clinical advice to the participants.

ELIGIBILITY:
Inclusion Criteria:

* Of age ≥18 years or older.
* Having a diagnosis of MM; newly diagnosed or relapsed/refractory disease
* Undergoing systemic treatment through the UAB MM Clinic Pathway
* Able to provide informed consent to be included in the intervention
* MM patients in a prior/concurrent (non-pyscho/educational intervention), MM study will be eligible to participate
* Have either SMS texting or email access to receive encouragement messages

Exclusion Criteria:

Patients will be ineligible for the program if they are:

* Being treated by end-of-life or comfort care measures only
* MM patients not treated through the UAB MM Clinic Pathway.
* MM patients not requiring systemic therapy.
* Patients with a diagnosis of MGUS or SMM.
* Have a history of other malignancy within the past [3 or 5] years with the exception of:
* Malignancies treated with curative intent and with no known active disease present for ≥ 3 (or 5) years before enrollment and felt to be at low risk for recurrence by the treating physician
* Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
* Adequately treated cervical carcinoma in situ without evidence of disease
* Adequately treated breast ductal carcinoma in situ without evidence of disease
* Prostatic intraepithelial neoplasia without evidence of prostate cancer
* Adequately treated urothelial papillary noninvasive carcinoma or carcinoma in situ
* Are enrolled in a prior/concurrent MM psycho-educational study

Other Exclusions:

* Patients who do not have either SMS texting or email access to receive encouragement messaging will be excluded
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
Assess baseline anxiety levels in MM patients undergoing therapy using the PROMIS assessment tool for anxiety | Baseline
  We will measure baseline anxiety levels in MM patients prior to implementation of educational program (MPI) using the PROMIS assessment tool for anxiety
Assess anxiety levels 12 weeks after educational program (MPI) in MM patients undergoing therapy using the PROMIS assessment tool for anxiety | 12 weeks post intervention
  We will measure anxiety levels in MM patients 12 weeks after implementation of educational program (MPI) using the PROMIS assessment tool for anxiety
Assess anxiety levels 24 weeks after educational program (MPI) in MM patients undergoing therapy using the PROMIS assessment tool for anxiety | 24 weeks post intervention
  We will measure anxiety levels in MM patients 24 weeks after implementation of educational program (MPI) using the PROMIS assessment tool for anxiety

SECONDARY OUTCOMES:
Assess baseline depression levels in MM patients using the PROMIS assessment tool for depression | Baseline
  We will measure baseline depression in MM patients prior to implementation of educational program using the PROMIS assessment tool for depression
Assess depression levels 12 weeks after education intervention (MPI) in MM patients using the PROMIS assessment tool for depression | 12 weeks post intervention
  We will assess outcomes 12 weeks after implementation of educational program using the PROMIS assessment tool for depression
Assess depression levels 24 weeks after education intervention (MPI) in MM patients using the PROMIS assessment tool for depression | 24 weeks post intervention
  We will assess outcomes 24 weeks after implementation of educational program using the PROMIS assessment tool for depression
Assess baseline patient self-efficacy for symptom management in MM patients using the PROMIS assessment tool for self-Efficacy | Baseline
  We will assess baseline patient self-efficacy for symptom management in MM patients before the implementation of educational program (MPI) using the PROMIS assessment tool for self-Efficacy
Assess patient self-efficacy for symptom management 12 weeks after educational program (MPI) in MM patients using the PROMIS assessment tool for self-Efficacy | 12 weeks post intervention
  We will assess outcomes 12 weeks after implementation of educational program (MPI) using the PROMIS assessment tool for self-Efficacy
Assess patient self-efficacy for symptom management 24 weeks after educational program (MPI) in MM patients using the PROMIS assessment tool for self-Efficacy | 24 weeks post intervention
  We will assess outcomes 24 weeks after implementation of educational program (MPI) using the PROMIS assessment tool for self-Efficacy
Assess baseline patient adherence to myeloma specific medication and treatment schedules in MM patients using the CASE Medication Adherence Index | Baseline
  We will baseline assess patient adherence to myeloma specific medication and treatment schedules in MM patients before the implementation of educational program (MPI) using the CASE Medication Adherence Index
Assess patient improvement in adherence to myeloma specific medication and treatment schedules 12 weeks after educational program (MPI) in MM patients using the CASE Medication Adherence Index | 12 weeks post intervention
  We will assess outcomes 12 weeks after implementation of educational program (MPI) using the CASE Medication Adherence Index
Assess patient improvement in adherence to myeloma specific medication and treatment schedules 24 weeks after educational program (MPI) in MM patients using the CASE Medication Adherence Index | 24 weeks post intervention
  We will assess outcomes 24 weeks after implementation of educational program (MPI) using the CASE Medication Adherence Index

OTHER OUTCOMES:
Assess baseline Qualityof Life (QoL) in MM patients undergoing therapy using EORTC-QLQ-C30, and FACIT-sp-12 questionnaires | Baseline
  We will baseline QoL in MM patients before implementation of educational program (MPI) using EORTC-QLQ-C30, and FACIT-sp-12 questionnaires
Assess effect on Qualityof Life (QoL) 12 weeks after educational program (MPI) in MM patients undergoing therapy using EORTC-QLQ-C30, and FACIT-sp-12 questionnaires | 12 weeks post intervention
  We will assess outcomes 12 weeks after implementation of educational program (MPI) using EORTC-QLQ-C30, and FACIT-sp-12 questionnaires
Assess effect on Qualityof Life (QoL) 24 weeks after educational program (MPI) in MM patients undergoing therapy using EORTC-QLQ-C30, and FACIT-sp-12 questionnaires | 24 weeks post intervention
  We will assess outcomes 24 weeks after implementation of educational program (MPI) using EORTC-QLQ-C30, and FACIT-sp-12 questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Smith Giri, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States